CLINICAL TRIAL: NCT00493363
Title: Clinical Investigation of In-vivo Susceptibility of P.Falciparum to Artesunate in Western Cambodia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: World Health Organization (Other); NCHADS - Ministry of Health of Cambodia (Other); Mahidol University (Other); Institut Pasteur (Industry); FHI 360 (Other); Li Ka Shing Foundation (Other)
Responsible Party: Principal Investigator, Arjen Dondorp, Deputy Director, University of Oxford
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-Dondorp
Record Dates: First submitted 2007-06-27; First posted 2007-06-28 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Falciparum Malaria
Keywords: falciparum malaria; artemisinins; artesunate; resistance
MeSH Terms: conditions — Malaria, Falciparum | interventions — Artesunate; Mefloquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- arm 1 (Experimental)
  Interventions: Drug: Artesunate
- arm 2 (Active Comparator)
  Interventions: Drug: Artesunate + Mefloquine

INTERVENTIONS:
Drug: Artesunate — Artesunate 2 mg/kg/day for 7 days
  Arms: arm 1
Drug: Artesunate + Mefloquine — Artesunate 4mg/kg/day for 3 days plus mefloquine 15mg/kg on day 3 and 10mg/kg on day 4
  Arms: arm 2

SUMMARY:
There are worrying signs that parasitological responses to the artemisinin drugs for uncomplicated falciparum malaria are slower than elsewhere in the world.If responses to artesunate are poor it is essential to have characterised the blood concentration profile as well as the parasitological response to differentiate resistance from abnormal pharmacokinetics.

The primary objective of the study is to assess the level of resistance to artemisinin derivatives in Western Cambodia.

A detailed evaluation of 2 different artesunate containing regimens in patients with uncomplicated malaria will be performed. Patients will be randomised to receive either a) Artesunate 2mg/kg/day for 7 days or b) Artesunate 4mg/kg/day for 3 days plus mefloquine 15mg/kg on day 3 and 10mg/kg on day 4 The effect on parasite clearance and cure will be assessed in relation to blood concentrations of the antimalarial drugs ('PK-PD').

DETAILED DESCRIPTION:
Primary objective:

To assess the level of resistance to artemisinin derivatives in Western Cambodia.

Secondary objective:

To assess the level of resistance to other antimalarial drugs in Western Cambodia

1. Background; There are worrying signs from Western Cambodia that parasitological responses to artesunate and artemether containing treatment regimens for uncomplicated falciparum malaria are slower than elsewhere in the world [1-4]. Both delayed parasite clearance and unusually high failure rates with artesunate-mefloquine and artemether-lumefantrine have been reported [1,2]. Although occasional poor responses to artesunate have been described previously [5] the current reports suggest a consistent problem. As the rate of parasite clearance is a good pharmacodynamic measure of efficacy of the artemisinin related compounds [6,7], this could indicate the emergence of significant resistance[8]. These antimalarials are central to current treatment strategies[9], and so spread of significant resistance outside this area would be a disaster. Radical containment measures might be needed. In this context there is an urgent need to proceed quickly to investigate the level of resistance to artemisinin derivatives in Western Cambodia to provide a definitive assessment so that if necessary containment plans can be developed in 2007. A group of malaria investigators from Cambodia and Thailand have joined together to address this urgent question as quickly and effectively as possible.

   The trial described here proposes to assess the current recommended doses given in the normal way, and if necessary a higher dose of artesunate. There is no known dose related toxicity with artesunate, and doses up to 10mg/kg/day have been given (by us) without any adverse effects[10]. The two features of this study which differ from normal studies in uncomplicated malaria are the repeated blood sampling and the 7 day in-patient stay. If responses to artesunate are poor it is essential to have characterised the blood concentration profile as well as the parasitological response to differentiate resistance from abnormal pharmacokinetics.
2. General Plan; The situation was reviewed in open forum by malaria experts from Cambodia, Thailand, and WHO, and was considered sufficiently worrying to prompt planning of an urgent investigation under the aegis of the Mekong Malaria Programme. First it is necessary to determine the level of in-vivo and in-vitro susceptibility to artemisinin derivatives. This will involve detailed clinical and laboratory studies associated with simultaneous assessment in-vitro in several laboratories including - A. National Malaria Control Programme, Pnomh Penh B. Mahidol Oxford Research Unit (MORU), Bangkok. C. Institut Pasteur, Pnomh Penh. D. Family Health International, Asia-Pacific Regional Office

   If artemisinin resistance is confirmed then
   1. plans for containment will need to be developed urgently.
   2. molecular genetic studies will be conducted to determine the basis of resistance.
   3. Epidemiological and behavioural studies will be conducted to inform how resistance may have been selected and how it might be contained

   This proposal describes the initial clinical studies which would be conducted by the Mahidol-University Research Unit, Bangkok together Family Health International under the leadership of the Cambodian NMCP. This will be an open randomised PK-PD comparison of artesunate versus artesunate-mefloquine.

   This clinical study will be conducted in Pailin, where poor parasitological responses to artesunate have been documented. FHI took on the management of a village malaria worker programme in Pailin, previously developed by MSF, and have developed the clinical facility. Trials of artesunate-pyronaridine, coordinated by FHI are now taking place there.

   2.1 Method A detailed pharmacokinetic-pharmacodynamic evaluation of artesunate in acute uncomplicated falciparum malaria will be conducted in Pailin Hospital.

   2.1.1.Timing Rainy season (May to December) 2007.

   2.1.2. Patients Children >5yrs and adults presenting with acute falciparum malaria (N=40) to Pailin hospital will be eligible for inclusion in this study provided that
   1. They or their parents/guardians give fully informed consent.
   2. They are not pregnant.
   3. They have not received antimalarial drugs in the previous 48 hours.
   4. P.falciparum parasitaemia exceeds 10,000/uL.
   5. Microscopy does not indicate a mixed infection.
   6. There is no history of allergy to artesunate or mefloquine.
   7. They agree to 7 days hospitalization.

   2.1.3. Recruitment, randomization and enrolment: Fever patients in the villages surrounding Pailin or in Pailin itself will be screened with a PfHRP2-based malaria rapid test (ParacheckR) by the village malaria workers. In case of a positive test result, the patient will be transported by the study team to Pailin Referral Hospital, where further consent and enrolment procedures will be conducted. It will be made clear from the outset that refusal to participate will in no way jeopardize subsequent antimalarial treatment.

   2.1.4.Patient information and remuneration The details of the study and the reason for the study will be explained in Khmer to the patients and relatives. It will be explained clearly that if the patient does not want to participate or continue with the study then this will not affect their treatment in any way. Patients will be recompensed for the stay in hospital and travel expenses for each outpatient visit at an appropriate local rate.

   If the patient fulfils the entry criteria and informed consent is obtained, the patient will be entered into the study. Basic demographic and clinical parameters, including blood pressure and pulse rate, respiratory rate, temperature, weight, spleen and liver size, will be entered into a case report form.

   2.1.5. Randomisation Computer-based randomisation will be balanced in previously prepared blocks of 10.

   2.1.6. 'Repeated dose' If the patient vomits within half an hour after intake of the antimalarial drugs, the dose will be repeated. If vomiting occurs between half and a whole hour, half of the dose will be repeated.

   2.1.7. 'Rescue treatment' If a patient develops signs of severe malaria, parenteral artesunate and parenteral quinine will be given in standard doses [9]. The combination is safe, and would be expected to be effective in case of high level artemisinin resistance [11]. If the patient has a less than 75% fall in parasitaemia by day 3 or has any persisting parasitaemia by day 7, he/she will require rescue treatment consisting of artesunate 6 mg/kg in combination with doxycycline 4 mg/kg for 7 days. In children below the age of 8, doxycycline should be replaced by clindamycin (10 mg/kg/dose, two times a day for 7 days)

   2.2. Procedures On enrollment a detailed history and full clinical examination will be performed and recorded on a standard CRF. Part of the blood sample will be taken at baseline for immediate culture (for an in-vitro susceptibility test) and also storage of parasites (cryopreserved in liquid nitrogen), parasite DNA and mRNA.

   2.2.1. Drugs Patients will be randomized to receive either
   1. Artesunate (Guilin Pharmaceutical Company, PRC) 2mg/kg/day for 7 days. N=20………………………………………………………………………….AS7
   2. Artesunate (Guilin Pharmaceutical Company, PRC) 4mg/kg/day for 3 days plus mefloquine 15mg/kg on day 3 and 10mg/kg on day 4 N=20………………………………………………………………………MAS3

   2.2.2. Blood collection on admission On admission blood will be collected for parasite count (thin and thick films stained by Field's method), CBC, and routine biochemistry. An additional 20 ml of blood will be collected in a sterile heparinised tube for parasite culture and cryopreservation, and 2 ml for assessment of drug levels (artesunate and mefloquine). The maximum volume taken from children < 10yrs is 10mL.

   2.2.4. Follow-up Patients will remain in hospital for 7 days or longer if parasites have not cleared. They will then be followed for 42 days and at each weekly visit will have a haematocrit and parasite count checked.

   2.3. Recurrent parasitaemia In case of recurrent falciparum malaria blood will be taken for cryopreserving parasites, antimalarial drug levels, for assessment of genotyping and gene expression (22mL). The maximum volume taken from children < 10yrs is 10mL. In case of recurrent parasitaemia, more than 3 days after the initiation of treatment, DNA will be isolated from from blood samples. Paired samples from every patient, taken at initial enrolment and at time of recurrence, will then be genotyped on the basis of polymorphisms in the genes for the merozoite surface proteins MSP-2 and MSP-1 and GLURP.
3. Measurements and analysis This is essentially a descriptive study so no formal sample size calculation is provided.

   3.1. Drug assays Artesunate, dihydroartemisinin and mefloquine will be measured in plasma samples. These assays will be performed in the MORU laboratories Bangkok.

   3.1.2. Analysis of PK data Conventional and population pharmacokinetic analyses will be performed (MORU). A PK-PD model will then be constructed. Artesunate and mefloquine will be characterized by conventional and population pharmacokinetic analyses.

   A population based pharmacokinetic-pharmacodynamic modelling approach will be used to describe the antimalarial effect of artesunate in patients with acute falciparum malaria. The objective of the modelling exercise is to characterise the relationship between pharmacokinetic variables and parasite clearance measures.

   The clinical and parasitological responses will be compared with previous data from Thailand and Cambodia.

   3.2 In-vitro testing On-site PfHRP2 based in-vitro testing will be performed . Parasites will be transported to Pnomh Penh and also cryopreserved for later testing.

   3.2.1. Molecular studies There will baseline genotyping as described above and also systematic screening for mixed infections. Putative resistance genes will be sequenced (e.g. PfATPase6) or copy number and expression assessed (PfMDR1).
4. Interim review and options for dose adjustment Monthly updates on recruitment and therapeutic responses will be provided to all participants from the study site.

   Artesunate should produce parasite reduction ratios of approximately 10,000/cycle, which result in parasite clearance times which are usually less than 48 hours. If six patients in either treatment group have PCTs >96 hours then the dosage of artesunate in that treatment arm will be increased AS7 2mg/kg/day increases to AS7 4mg/kg/day MAS3 4mg/kg/day increases to MAS3 6mg/kg/day The sample size will be reviewed at this time.
5. Treatment of recurrent falciparum malaria infections Patients with recurrent infections will receive an increased dose of artesunate in the retreatment.

Recurrent infections following the 7 day regimen will receive artesunate 4 mg/kg/day for 7 days. Recurrences following the MAS3 regimen will receive artesunate 6 mg/kg/day for 7 days Children aged over 8 years will receive doxycycline 200mg day in addition, and those between 6 and 8 will receive clindamycin 10mg/kg bid Patients with recrudescences will be restudied as above provided they agree.

ELIGIBILITY:
Inclusion Criteria:

* Children >5yrs and adults presenting with acute falciparum malaria (N=40) to Pailin hospital will be eligible for inclusion in this study provided that

  * They or their parents/guardians give fully informed consent.
  * They are not pregnant.
  * They have not received antimalarial drugs in the previous 48 hours.
  * P.falciparum parasitaemia exceeds 10,000/uL

Exclusion Criteria:

* Mixed infection (such as vivax malaria), history of allergy to artesunate or mefloquine, any sign of severe disease according to WHO criteria

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
parasite clearance times in relation to artesunate/DHA plasma concentrations (PK-PD) | June 2008
  parasite clearance times in relation to artesunate/DHA plasma concentrations (PK-PD)

SECONDARY OUTCOMES:
56 day cure rates, in vitro sensitivity, molecular markers of drug resistance | June 2008
  56 day cure rates, in vitro sensitivity, molecular markers of drug resistance

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas J White, DSc,FRCP,FRS, Principal Investigator — Oxford University/ Mahidol University; Duong Socheat, MD, Study Chair — National Malaria Control Programme Cambodia
Locations (1):
- Pailin Referal Hospital, Pailin, Cambodia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mechri M, Epaud R, Emond S, Coulomb A, Jaubert F, Tarrant A, Feldmann D, Flamein F, Clement A, de Blic J, Taam RA, Brunelle F, le Pointe HD. Surfactant protein C gene (SFTPC) mutation-associated lung disease: high-resolution computed tomography (HRCT) findings and its relation to histological analysis. Pediatr Pulmonol. 2010 Oct;45(10):1021-9. doi: 10.1002/ppul.21289. PMID 20658481
- [Derived] Anderson TJ, Nair S, Nkhoma S, Williams JT, Imwong M, Yi P, Socheat D, Das D, Chotivanich K, Day NP, White NJ, Dondorp AM. High heritability of malaria parasite clearance rate indicates a genetic basis for artemisinin resistance in western Cambodia. J Infect Dis. 2010 May 1;201(9):1326-30. doi: 10.1086/651562. PMID 20350192
- [Derived] Dondorp AM, Nosten F, Yi P, Das D, Phyo AP, Tarning J, Lwin KM, Ariey F, Hanpithakpong W, Lee SJ, Ringwald P, Silamut K, Imwong M, Chotivanich K, Lim P, Herdman T, An SS, Yeung S, Singhasivanon P, Day NP, Lindegardh N, Socheat D, White NJ. Artemisinin resistance in Plasmodium falciparum malaria. N Engl J Med. 2009 Jul 30;361(5):455-67. doi: 10.1056/NEJMoa0808859. PMID 19641202